CLINICAL TRIAL: NCT02544048
Title: Markers of T Cell Suppression: Antimalarial Treatment and Vaccine Responses in Healthy Malian Adults
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999915197; 15-I-N197
Record Dates: First submitted 2015-09-05; First posted 2015-09-09 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2017-08-11

CONDITIONS: Malaria
Keywords: Immune; Parasitemia; Menactra; Polymerase Chain Reaction (PCR); Coartem
MeSH Terms: conditions — Malaria; Parasitemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Background:

People with malaria often show altered immune responses to many illnesses and vaccines. This means that the malaria might cause immune suppression. It is not clear how or which vaccines are impacted by malaria. It is also not clear if the impacts are such that people should be preemptively treated before they get vaccinations. Researchers want to see if there is a link between taking an antimalaria drug prior to getting vaccines and the immune response to those vaccines. To do this, they will study people who are taking part in certain NIAID studies.

Objectives:

To compare the proportion of PD1+ CD4 T cells among all T cells in vaccine immune responses in adults who have or have not received antimalarials prior to getting a Menactra vaccine.

Eligibility:

Healthy Malian adults who:

Were previously enrolled in NIAID Protocol 13-I-N109 or 15-I-0044

Reside in Bancoumana and neighboring villages

Are not pregnant

Design:

Participants will be screened with a physical exam.

Participants will get the vaccines listed below as part of Protocol 13-I-N109 or 15-I-0044. This study will follow their schedule.

At each visit, participants will give a blood sample. They will also have a physical exam. Each visit will last 1 to 2 hours.

At visit 1, participants will get a hepatitis vaccine.

Two weeks later, participants may get the antimalarial drug Coartem . They will be chosen at random.

Two weeks later, participants will get Menactra .

Participants will have 5 follow-up visits after they get Menactra .

The study will last up to 4 months.

...

DETAILED DESCRIPTION:
Malaria patients often show altered immune responses, not only to malaria parasites but also to unrelated pathogens (eg, HIV, EBV, salmonella, helminthes) and antigens, including routine vaccines, suggesting that there is an active immune suppression or more accurately perhaps, immunomodulation, occurring during the course of malaria infection. How and which vaccines are impacted by clinical malaria or asymptomatic parasitemia is not completely clear and nor is whether the impacts are significant enough to recommend delaying or pre-emptively treating individuals prior to vaccinations.

Up to 75 adults will be recruited from volunteers enrolled in NIAID protocol 13-I-N109 and NIAID protocol 15-I-0044 who after unblinding have opted to receive or complete the comparator vaccine series: Euvax (Hepatitis B) or TWINRIX (Hepatitis B) and Menactra (Meningococcal). This longitudinal study will be conducted in Bancoumana and neighboring villages in Mali. In September 2015, up to 50 adults presenting for their Vaccination #3 of Euvax will be enrolled from NIAID protocol 13-I-N109. In October 2015, up to 25 adults presenting for their Study Day 168 will be enrolled following unblinding from NIAID protocol 15-I-0044.

Following receipt of their Euvax B or TWINRIX vaccination, subjects will be randomized to receive or not receive a course of Coartem (artemether-lumefantrine) 2 weeks prior to their scheduled Menactra vaccination. They will then be followed for approximately 3 months post receipt of Menactra . Samples will be collected from the adults at the time of prior to and following receipt of both vaccinations and assessed in ex vivo assays for markers of T-cell suppression as the primary outcome of this study. For our secondary outcomes, we will examine levels of regulatory T cells, measure T cell responses in stimulation assays, and survey parasitemia by blood smear and by polymerase chain reaction assays. We expect that levels of T-cell suppression and regulatory T cells will be similar between groups before antimalarial treatment or malaria infection, but after treatment or in those subjects that remain uninfected these levels will be significantly lower as compared to the untreated and or infected subjects.

ELIGIBILITY:
* INCLUSION
* Enrolled, completed unblinding, and have opted to receive the comparator vaccines in either NIAID Protocol 13-I-N109 or 15-I-0044
* In good general health and without any clinically significant medical history
* Willing to have blood samples stored for future research
* Known resident of Bancoumana or surrounding area

EXCLUSION

* Known to be pregnant (by history)
* Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, endocrine, rheumatologic, autoimmune, hematological, oncologic, psychiatric, or renal disease by history and/or physical examination
* Behavioral, cognitive, or psychiatric disease that in the opinion of the investigator affects the ability of the participant to understand and comply with the study protocol
* Prior to Study Day 0, receipt of a live vaccine within the past 4 weeks or a killed vaccine within the past 2 weeks
* Use of chronic (greater than or equal to 14 days) oral or intravenous corticosteroids (excluding topical or nasal) at immunosuppressive doses (eg, prednisone > 10 mg/day) or immunosuppressive drugs within 30 days of Study Day 0
* Known allergies or contraindications to study treatment (Coartem [artemether//lumefantrine]) or vaccines (Euvax B or TWINRIX and Menactra )
* Other condition that in the opinion of the investigator would jeopardize the safety or rights of a participant participating in the trial, interfere with the evaluation of the study objectives, or would render the subject unable to comply with the protocol

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2015-09-04; Primary Completion 2015-09-04 (Actual); Study Completion 2017-08-11 (Actual)

PRIMARY OUTCOMES:
Proportion of T cells expressing PD-1 among all T cells on Study Day 42 | Study Day 42

CONTACTS AND LOCATIONS:
Overall Officials: Sara A Healy, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- Malaria Research and Training Center, Bamako, Mali

REFERENCES:
- [Background] Williamson WA, Greenwood BM. Impairment of the immune response to vaccination after acute malaria. Lancet. 1978 Jun 24;1(8078):1328-9. doi: 10.1016/s0140-6736(78)92403-0. PMID 78096
- [Background] Cunnington AJ, Riley EM. Suppression of vaccine responses by malaria: insignificant or overlooked? Expert Rev Vaccines. 2010 Apr;9(4):409-29. doi: 10.1586/erv.10.16. PMID 20370551
- [Background] Greenwood BM, Bradley-Moore AM, Bryceson AD, Palit A. Immunosuppression in children with malaria. Lancet. 1972 Jan 22;1(7743):169-72. doi: 10.1016/s0140-6736(72)90569-7. No abstract available. PMID 4109547